CLINICAL TRIAL: NCT01897571
Title: An Open-Label, Multicenter, Phase 1/2 Study of Tazemetostat as a Single Agent in Subjects With Advanced Solid Tumors or With B-cell Lymphomas and Tazemetostat in Combination With Prednisolone in Subjects With Diffuse Large B Cell Lymphoma
Brief Title: Study of Tazemetostat as Single Agent in Solid Tumors or B-cell Lymphomas and in Combination With Prednisolone in DLBCL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7438-G000-101; 2012-004083-21 (EudraCT Number)
Record Dates: First submitted 2013-06-21; First posted 2013-07-12 (Estimated); Results first posted 2023-08-04 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: B-cell Lymphomas (Phase 1); Advanced Solid Tumors (Phase 1); Diffuse Large B-cell Lymphoma (Phase 2); Follicular Lymphoma (Phase 2); Transformed Follicular Lymphoma; Primary Mediastinal Large B-Cell Lymphoma
Keywords: Epizyme; Tazverik; Tazemetostat (EPZ-6438)
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — tazemetostat; Prednisolone; prednisolone phosphate; Methylprednisolone; prednisolone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 (Experimental): Patients in the Phase 1 portion of the study.
  Interventions: Drug: Tazemetostat
- Phase 2 Group 1: Tazemetostat in R/R FL with Mutant EZH2 (Experimental): Patients with R/R FL with mutant EZH2 treated with tazemetostat as a single agent in Phase 2 of the study.
  Interventions: Drug: Tazemetostat
- Phase 2 Group 2: Tazemetostat in R/R FL with Wild-Type EZH2 (Experimental): Patients with R/R FL with wild-type EZH2 treated with tazemetostat as a single agent in Phase 2 of the study.
  Interventions: Drug: Tazemetostat
- Phase 2 Group 3: Tazemetostat in R/R DLBCL (Experimental): Patients with R/R DLBCL treated with tazemetostat as a single agent or tazemetostat in combination with prednisolone in Phase 2 of the study.
  Interventions: Drug: Tazemetostat; Drug: Prednisolone

INTERVENTIONS:
Drug: Tazemetostat — Patients who received 800 mg of tazemetostat, BID, administered in continuous 28-day cycles.
  Other Names: EPZ-6438; E7438
  Arms: Phase 2 Group 1: Tazemetostat in R/R FL with Mutant EZH2; Phase 2 Group 2: Tazemetostat in R/R FL with Wild-Type EZH2; Phase 2 Group 3: Tazemetostat in R/R DLBCL
Drug: Prednisolone — Patients who received 40 mg/m^2 prednisolone once daily on Days 1-5 and 15-19 of Cycles 1-4.
  Other Names: Pediapred; Omnipred; Pred Mild; Pred Forte,; Orapred ODT,; Veripred 20,; Millipred DP
  Arms: Phase 2 Group 3: Tazemetostat in R/R DLBCL
Drug: Tazemetostat — Patients who received 100 mg to 1600 mg of tazemetostat, BID, administered in continuous 28-day cycles.
  Other Names: EPZ-6438; E7438
  Arms: Phase 1

SUMMARY:
This is an open-label, multicenter, Phase 1/2 study of tazemetostat as a single agent in subjects with advanced solid tumors or with B-cell lymphomas and tazemetostat in combination with prednisolone in subjects with diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase 1/2 study conducted in two parts: The Phase 1 part comprised dose escalation and expansion to establish the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) when tazemetostat was given twice daily (BID) orally on a continuous basis. Additionally, in separate cohorts in Phase 1, the effect of food on the bioavailability of tazemetostat as well as the drug-drug interaction (DDI) potential of tazemetostat were evaluated. The Phase 2 part was initiated once the RP2D was established. Phase 2 enrolled subjects with relapsed/ refectory (R/R) DLBCL (Cohorts 1-3 and 6) and subjects with R/R FL (Cohorts 4 and 5) for the determination of efficacy and safety of tazemetostat monotherapy (Cohorts 1-5) and of tazemetostat in combination with prednisolone (Cohort 6) with placement determined by centrally confirmed histology, cell of origin (COO), and enhancer of zeste homologue 2 (EZH2) mutation status.

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1: Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Phase 2: ECOG performance status of 0 to 2.
2. Life expectancy of at least 3 months before starting tazemetostat.
3. Voluntary agreement to provide written informed consent and willing to adhere to all protocol requirements
4. Subjects with Hepatitis B or C are eligible on the condition that subjects have adequate liver function and are hepatitis B surface antigen negative and/or have undetectable hepatitis C virus (HCV) RNA.
5. Adequate renal and liver function
6. Phase 1: Males or females aged ≥ 16 years at time of informed consent. Phase 2: Males or females aged ≥ 18 years at the time of informed consent .
7. Females must not be lactating or pregnant at screening or baseline as documented by a negative pregnancy test All females will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months consecutive amenorrheic, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least 1 month before dose). Females of childbearing potential must not have had unprotected sexual intercourse within 30 days prior to study entry and must agree to use a highly effective method of contraception, from the last menstrual period prior to randomization, during Treatment Cycles, and for 6 months after the last final dose of study drug; any male partner must use a condom.
8. Male subjects must have had a successful vasectomy (with confirmed azoospermia) or they and their female partner must meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception and use a condom throughout the study period and for 3 months after study drug discontinuation). Nonvasectomized male subjects must also agree to refrain from donating sperm from first dose of tazemetostat until 3 months following the last dose of tazemetostat
9. Phase 1 only: Histologically and/or cytologically confirmed advanced or metastatic solid tumor or B-cell lymphomas that have progressed after treatment with approved therapies or for which there are no standard therapies available.
10. Phase 2, Groups 1-6 only: Subjects must satisfy all of the following criteria:

    1. Have histologically confirmed DLBCL (including primary mediastinal B-cell lymphoma), with relapsed or refractory disease following at least 2 lines of prior standard therapy, including alkylator/anthracycline (unless anthracycline-based chemotherapy is contraindicated)/anti-CD20-based therapy (rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone [R-CHOP] or equivalent) AND must be considered unable to benefit from intensification treatment with autologous hematopoietic stem cell transplantation (ASCT) as defined by meeting at least 1 of the following criteria:

       * Relapsed following, or refractory to, previous ASCT
       * Did not achieve at least a partial response to a standard salvage regimen (eg, rituximab, ifosfamide, carboplatin, and etoposide phosphate [R-ICE] or rituximab, dexamethasone, cytarabine, and cisplatin [R-DHAP])
       * Ineligible for intensification treatment due to age or significant comorbidity
       * Ineligible for intensification treatment due to failure to mobilize an acceptable number of hematopoietic stem cells
       * Refused intensification treatment and/or ASCT or
    2. Have histologically confirmed Follicular Lymphoma (FL), all grades. Subjects may have relapsed/refractory disease following at least 2 standard prior systemic treatment regimens where at least 1 anti-CD20-based regimen was used. Subjects with prior radiotherapy will be included; however, radiotherapy alone will not be considered a systemic treatment regimen.
    3. Have provided sufficient archival tumor tissue that has been successfully tested for EZH2 mutation status and cell of origin (DLBCL only)
    4. Have measurable disease as defined by International Working Group-Non-Hodgkin's Lymphoma (IWG-NHL)

Exclusion Criteria:

1. Prior exposure to tazemetostat or other inhibitor(s) of EZH2.
2. Subjects with leptomeningeal metastases or brain metastases or history of previously treated brain metastases.
3. Has thrombocytopenia, neutropenia, or anemia of Grade ≥3 (per CTCAE 4.03 criteria) and any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS).
4. Has a prior history of T-cell lymphoblastic lymphoma(T-LBL) or T-cell lymphoblastic leukemia (T-ALL).
5. Subjects taking medications that are known strong CYP3A inhibitors and strong or moderate CYP3A inducers (including St. Johns Wort) 6. Subjects unwilling to remove Seville oranges, grapefruit juice and grapefruit from their diet.
6. Any unstable or unresolved prior treatment-related (i.e. chemotherapy, immunotherapy, radiotherapy) toxicities at time of enrollment.
7. Major surgery within 4 weeks before the first dose of study drug. .
8. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the bioavailability of tazemetostat.
9. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug; or cardiac ventricular arrhythmia.
10. Venous thrombosis or pulmonary embolism within the last 3 months before starting tazemetostat.
11. Active infection requiring systemic therapy.
12. Immunocompromised patients, including patients known to be infected with human immunodeficiency virus (HIV).
13. Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study.
14. Females who are pregnant or breastfeeding.
15. Phase 2 only: Subjects with noncutaneous malignancies other than B-cell lymphomas. Exception: Subjects with another malignancy who have been disease-free for 5 years, or subjects with a history of a completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-06-13 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (52):
- United States (12):
  - Birmingham, Alabama
  - Duarte, California
  - Santa Barbara, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Ocala, Florida
  - Ann Arbor, Michigan
  - New York, New York
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Seattle, Washington
- Australia (3):
  - Clayton
  - Geelong
  - Melbourne
- Canada (2):
  - Montreal
  - Toronto
- France (13):
  - Bordeaux
  - Caen
  - Créteil
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Pierre-Bénite
  - Rennes
  - Rouen
  - Villejuif
- Germany (2):
  - Göttingen
  - Münster
- Italy (2):
  - Bologna
  - Napoli
- Poland (4):
  - Krakow
  - Lublin
  - Poznan
  - Warsaw
- Taipei, Taiwan
- Ukraine (9):
  - Chernivtsi
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Mykolayiv
  - Uzhhorod
  - Zaporizhzhya
  - Zhytomyr
- United Kingdom (4):
  - Glasgow
  - London
  - Manchester
  - Southampton

REFERENCES:
- [Derived] Alfaifi A, Bahashwan S, Alsaadi M, Ageel AH, Ahmed HH, Fatima K, Malhan H, Qadri I, Almehdar H. Advancements in B-Cell Non-Hodgkin's Lymphoma: From Signaling Pathways to Targeted Therapies. Adv Hematol. 2024 Nov 12;2024:5948170. doi: 10.1155/2024/5948170. eCollection 2024. PMID 39563886
- [Derived] Bosch F, Kuruvilla J, Vassilakopoulos TP, Maio DD, Wei MC, Zumofen MB, Nastoupil LJ. Indirect Treatment Comparisons of Mosunetuzumab With Third- and Later-Line Treatments for Relapsed/Refractory Follicular Lymphoma. Clin Lymphoma Myeloma Leuk. 2024 Feb;24(2):105-121. doi: 10.1016/j.clml.2023.09.007. Epub 2023 Sep 28. PMID 37981564
- [Derived] Morschhauser F, Tilly H, Chaidos A, McKay P, Phillips T, Assouline S, Batlevi CL, Campbell P, Ribrag V, Damaj GL, Dickinson M, Jurczak W, Kazmierczak M, Opat S, Radford J, Schmitt A, Yang J, Whalen J, Agarwal S, Adib D, Salles G. Tazemetostat for patients with relapsed or refractory follicular lymphoma: an open-label, single-arm, multicentre, phase 2 trial. Lancet Oncol. 2020 Nov;21(11):1433-1442. doi: 10.1016/S1470-2045(20)30441-1. Epub 2020 Oct 6. PMID 33035457
- [Derived] Italiano A, Soria JC, Toulmonde M, Michot JM, Lucchesi C, Varga A, Coindre JM, Blakemore SJ, Clawson A, Suttle B, McDonald AA, Woodruff M, Ribich S, Hedrick E, Keilhack H, Thomson B, Owa T, Copeland RA, Ho PTC, Ribrag V. Tazemetostat, an EZH2 inhibitor, in relapsed or refractory B-cell non-Hodgkin lymphoma and advanced solid tumours: a first-in-human, open-label, phase 1 study. Lancet Oncol. 2018 May;19(5):649-659. doi: 10.1016/S1470-2045(18)30145-1. Epub 2018 Apr 9. PMID 29650362

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Tazemetostat 100 mg: Patients received tazemetostat 100 milligrams (mg) tablets orally twice daily (BID) in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 1: Tazemetostat 200 mg: Patients received tazemetostat 200 mg tablets orally BID in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 1: Tazemetostat 400 mg: Patients received tazemetostat 400 mg tablets orally BID in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 1: Tazemetostat 800 mg: Patients received tazemetostat 800 mg tablets orally BID in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 1: Tazemetostat 1600 mg: Patients received tazemetostat 1600 mg tablets orally BID in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 1: Food Effect (All Patients): Patients received tazemetostat 200 mg as a single oral dose on Day -8 either after fasting for 8 hours before dosing or immediately after consuming a high-fat breakfast on Day -8. Following a 7-day washout period, patients crossed over to receive the second tazemetostat 200 mg single oral dose on Day -1 in the opposite condition (fed or fasted).
- Phase 1: Tazemetostat 800 mg + Midazolam 2 mg: Patients received tazemetostat 800 mg orally BID continuously starting on Day 1, with a single oral dose of midazolam 2 mg administered on Day -1 and then on Day 15. Post Day 15, patients continued to receive tazemetostat 800 mg tablets orally BID in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 2 Group 1: Tazemetostat in Relapsed/Refractory (R/R) Follicular Lymphoma (FL) With Mutant EZH2: Patients with R/R FL with mutant enhancer of zeste homolog 2 (EZH2) treated with tazemetostat as a single agent in Phase 2 of the study. Patients received 800 mg of tazemetostat, orally BID, administered in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 2 Group 2: Tazemetostat in R/R FL With Wild-Type EZH2: Patients with R/R FL with wild-type EZH2 treated with tazemetostat as a single agent in Phase 2 of the study. Patients received 800 mg of tazemetostat, orally BID, administered in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 2 Group 3: Tazemetostat in R/R Diffuse Large B-cell Lymphoma (DLBCL) Monotherapy: Patients with R/R DLBCL received 800 mg of tazemetostat monotherapy, orally BID, administered in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 2 Group 4: Tazemetostat + Prednisolone in R/R DLBCL Combination Therapy: Patients received tazemetostat 800 mg tablets orally BID in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent. In addition, these patients also received prednisolone 40 mg/meter square (m^2) on Days 1 to 5 and 15 to 19 from Cycle 1 to Cycle 4 post which tazemetostat monotherapy was continued.
Period: Overall Study
Arm/Group | Phase 1: Tazemetostat 100 mg | Phase 1: Tazemetostat 200 mg | Phase 1: Tazemetostat 400 mg | Phase 1: Tazemetostat 800 mg | Phase 1: Tazemetostat 1600 mg | Phase 1: Food Effect (All Patients) | Phase 1: Tazemetostat 800 mg + Midazolam 2 mg | Phase 2 Group 1: Tazemetostat in Relapsed/Refractory (R/R) Follicular Lymphoma (FL) With Mutant EZH2 | Phase 2 Group 2: Tazemetostat in R/R FL With Wild-Type EZH2 | Phase 2 Group 3: Tazemetostat in R/R Diffuse Large B-cell Lymphoma (DLBCL) Monotherapy | Phase 2 Group 4: Tazemetostat + Prednisolone in R/R DLBCL Combination Therapy
Started | 6 | 3 | 3 | 14 | 12 | 13 | 13 | 48 | 54 | 163 | 71
Completed | 0 | 1 | 0 | 5 | 0 | 0 | 1 | 16 | 19 | 20 | 6
Not Completed | 6 | 2 | 3 | 9 | 12 | 13 | 12 | 32 | 35 | 143 | 65
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 1
Not completed — Other | 1 | 0 | 0 | 3 | 3 | 4 | 7 | 0 | 0 | 0 | 0
Not completed — Enrolled in rollover study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 7 | 9 | 1
Not completed — Death | 2 | 2 | 3 | 6 | 7 | 9 | 5 | 22 | 23 | 129 | 59

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Tazemetostat 100 mg: Patients received tazemetostat 100 mg tablets orally BID in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 2 Group 1: Tazemetostat in R/R FL With Mutant EZH2: Patients with R/R FL with mutant EZH2 treated with tazemetostat as a single agent in Phase 2 of the study. Patients received 800 mg of tazemetostat, orally BID, administered in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
  Tazemetostat: Patients who received 800 mg of tazemetostat, BID, administered in continuous 28-day cycles.
- Phase 2 Group 3: Tazemetostat in R/R DLBCL Monotherapy: Patients with R/R DLBCL received 800 mg of tazemetostat monotherapy, orally BID, administered in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
  Tazemetostat: Patients who received 800 mg of tazemetostat, BID, administered in continuous 28-day cycles.
- Phase 2 Group 4: Tazemetostat + Prednisolone in R/R DLBCL Combination Therapy: Patients received tazemetostat 800 mg tablets orally BID in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent. In addition, these patients also received prednisolone 40 mg/m^2 on Days 1 to 5 and 15 to 19 from Cycle 1 to Cycle 4 post which tazemetostat monotherapy was continued.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Tazemetostat 100 mg | Phase 1: Tazemetostat 200 mg | Phase 1: Tazemetostat 400 mg | Phase 1: Tazemetostat 800 mg | Phase 1: Tazemetostat 1600 mg | Phase 1: Food Effect (All Patients) | Phase 1: Tazemetostat 800 mg + Midazolam 2 mg | Phase 2 Group 1: Tazemetostat in R/R FL With Mutant EZH2 | Phase 2 Group 2: Tazemetostat in R/R FL With Wild-Type EZH2 | Phase 2 Group 3: Tazemetostat in R/R DLBCL Monotherapy | Phase 2 Group 4: Tazemetostat + Prednisolone in R/R DLBCL Combination Therapy | Total
Number analyzed (Participants) | 6 | 3 | 3 | 14 | 12 | 13 | 13 | 48 | 54 | 163 | 71 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (15.74) | 55.0 (30.20) | 59.0 (7.00) | 56.4 (13.54) | 51.6 (21.42) | 53.2 (16.39) | 55.0 (13.66) | 62.0 (8.83) | 61.1 (11.38) | 63.2 (14.35) | 65.4 (11.78) | 61.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 4 | 5 | 7 | 8 | 26 | 20 | 72 | 32 | 176
  Male | 5 | 2 | 3 | 10 | 7 | 6 | 5 | 22 | 34 | 91 | 39 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 7
  Not Hispanic or Latino | 2 | 1 | 2 | 7 | 6 | 10 | 11 | 38 | 26 | 103 | 62 | 268
  Unknown or Not Reported | 4 | 2 | 1 | 7 | 6 | 3 | 2 | 10 | 25 | 57 | 8 | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 2 | 1 | 2 | 7 | 6 | 10 | 11 | 33 | 15 | 71 | 28 | 186
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 1 | 7 | 6 | 3 | 2 | 15 | 38 | 89 | 41 | 208

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Tazemetostat as a Single-Agent and in Combination With Prednisolone (Phase 1 Only)
Description: Recommended Phase 2 dose (RP2D) of tazemetostat as administered orally twice daily (BID), continuously in 28-day cycles in subjects with advanced solid tumors or with relapsed and/or refractory B cell lymphomas as determined by incidence, seriousness, toxicity grade, and relatedness of treatment emergent dose limiting toxicities
Time Frame: The first 28-day cycle of therapy
Measure: Number; unit: mg BID
Groups:
- Phase 1: Patients in the Phase 1 portion of the study. Tazemetostat: Patients who received 100 mg to 1600 mg of tazemetostat, BID, administered in continuous 28-day cycles.
Arm/Group | Phase 1
Number analyzed (Participants) | 64
mg BID | 800

2. Primary Outcome: Objective Response Rate (ORR; Complete Response + Partial Response [CR + PR]) (Phase 2)
Description: Number of patients achieving an objective response (CR or PR)/number of patients treated x 100%. ORR was calculated as the percentage of patients with a confirmed complete response (CR) or partial response (PR) relative to the total number of patients in the analysis population per response evaluation criteria in solid tumors (RECIST) version (v)1.1. Complete Response (CR) was defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Radiologic tumor assessments performed at baseline(within 28 days before start of study treatment)and every 8 weeks during Cycles 2 to 6,and then every 12 weeks thereafter until confirmed disease progression (PD)/death,a maximum of approximately 82 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 Group 1: Tazemetostat in R/R FL With Mutant EZH2: Patients with R/R FL with mutant EZH2 treated with tazemetostat as a single agent in Phase 2 of the study. Patients received 800 mg of tazemetostat, orally BID, administered in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
- Phase 2 Group 3: Tazemetostat in R/R DLBCL Monotherapy: Patients with R/R DLBCL received 800 mg of tazemetostat monotherapy, orally BID, administered in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent.
Arm/Group | Phase 2 Group 1: Tazemetostat in R/R FL With Mutant EZH2 | Phase 2 Group 2: Tazemetostat in R/R FL With Wild-Type EZH2 | Phase 2 Group 3: Tazemetostat in R/R DLBCL Monotherapy | Phase 2 Group 4: Tazemetostat + Prednisolone in R/R DLBCL Combination Therapy
Number analyzed (Participants) | 48 | 54 | 163 | 71
Participants | 34 | 19 | 30 | 8

3. Secondary Outcome: Duration of Response for Tazemetostat as a Single Agent or in Combination With Prednisolone (Phase 2 Only)
Description: The time (in months) from the date of the initial response (CR or PR, whichever was first) until the date of the first documented disease progression per an Independent Review Committee (for Groups 1 and 2), per Investigator (Group 3), or death due to any cause. Patients who were alive and progression free at the time of the analysis were censored at the last date where the patient was known to be in response. Note: the DOR was censored, meaning data collection was stopped early for analysis, making the top limit of the 95% confidence interval not estimable (NE). Per RECIST v.1.0, CR was defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 mm in the short axis. The PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Radiologic tumor assessments performed at baseline (within 28 days before start of study treatment) and every 8 weeks during Cycles 2 to 6, and then every 12 weeks thereafter until confirmed PD/death, a maximum of approximately 82 months
Population: Patients who had a complete or partial response per an Independent Review Committee. Note: the DOR for some patients was censored, meaning data collection was stopped early for analysis making the top limit of the 95% confidence interval not estimable.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2 Group 4: Tazemetostat + Prednisone in R/R DLBCL Combination Therapy: Patients received tazemetostat 800 mg tablets orally BID in continuous 28-day treatment cycles until confirmed disease progression, unacceptable toxicity, or withdrawal of consent. In addition, these patients also received prednisolone 40 mg/m^2 on Days 1 to 5 and 15 to 19 from Cycle 1 to Cycle 4 post which tazemetostat monotherapy was continued.
Arm/Group | Phase 2 Group 1: Tazemetostat in R/R FL With Mutant EZH2 | Phase 2 Group 2: Tazemetostat in R/R FL With Wild-Type EZH2 | Phase 2 Group 3: Tazemetostat in R/R DLBCL Monotherapy | Phase 2 Group 4: Tazemetostat + Prednisone in R/R DLBCL Combination Therapy
Number analyzed (Participants) | 34 | 19 | 163 | 71
months | 11.3 [7.2 to NA] — NA indicates that upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events at study closure. | 13.0 [5.6 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | 5.8 [3.7 to 12.8] | 5.7 [2.1 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at study closure.

4. Secondary Outcome: Progression Free Survival for Tazemetostat as a Single Agent or in Combination With Prednisolone (Phase 2 Only)
Description: The time (in months) from the date of first dose of tazemetostat until the earliest date of disease progression or death from any cause. Per RECIST v1.0, CR was defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 mm in the short axis. The PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: as for outcome 3
Population: Patients who had a response event per Independent Review Committee.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Group 1: Tazemetostat in R/R FL With Mutant EZH2 | Phase 2 Group 2: Tazemetostat in R/R FL With Wild-Type EZH2 | Phase 2 Group 3: Tazemetostat in R/R DLBCL Monotherapy | Phase 2 Group 4: Tazemetostat + Prednisolone in R/R DLBCL Combination Therapy
Number analyzed (Participants) | 48 | 54 | 163 | 71
months | 13.8 [10.9 to 22.1] | 11.1 [3.7 to 14.6] | 1.9 [1.8 to 3.2] | 1.8 [1.6 to 2.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are reported from the first dose of study drug (Day 1) until confirmed disease progression, unacceptable toxicity, or withdrawal of consent. A maximum of approximately 40 months for Phase 1 and 82 months for Phase 2
Description: The safety population included all patients in the Intent-to-treat (ITT) population set who had at least 1 post-dose safety observation recorded. MedDRA v17.1 for Phase 1 and MedDRA v18.1 for Phase 2.
Arm/Group | Phase 1: Tazemetostat 100 mg | Phase 1: Tazemetostat 200 mg | Phase 1: Tazemetostat 400 mg | Phase 1: Tazemetostat 800 mg | Phase 1: Tazemetostat 1600 mg | Phase 1: Food Effect (All Patients) | Phase 1: Tazemetostat 800 mg + Midazolam 2 mg | Phase 2 Group 1: Tazemetostat in R/R FL With Mutant EZH2 | Phase 2 Group 2: Tazemetostat in R/R FL With Wild-Type EZH2 | Phase 2 Group 3: Tazemetostat in R/R DLBCL Monotherapy | Phase 2 Group 4: Tazemetostat + Prednisolone in R/R DLBCL Combination Therapy
All-Cause Mortality (participants affected / at risk) | 2/6 | 2/3 | 3/3 | 6/14 | 7/12 | 9/13 | 5/13 | 22/48 | 23/54 | 129/163 | 59/71
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/3 | 2/3 | 2/14 | 5/12 | 6/13 | 2/13 | 14/48 | 16/54 | 84/163 | 47/71
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 12/14 | 11/12 | 12/13 | 13/13 | 46/48 | 53/54 | 147/163 | 56/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Tazemetostat 100 mg (N=6) | Phase 1: Tazemetostat 200 mg (N=3) | Phase 1: Tazemetostat 400 mg (N=3) | Phase 1: Tazemetostat 800 mg (N=14) | Phase 1: Tazemetostat 1600 mg (N=12) | Phase 1: Food Effect (All Patients) (N=13) | Phase 1: Tazemetostat 800 mg + Midazolam 2 mg (N=13) | Phase 2 Group 1: Tazemetostat in R/R FL With Mutant EZH2 (N=48) | Phase 2 Group 2: Tazemetostat in R/R FL With Wild-Type EZH2 (N=54) | Phase 2 Group 3: Tazemetostat in R/R DLBCL Monotherapy (N=163) | Phase 2 Group 4: Tazemetostat + Prednisolone in R/R DLBCL Combination Therapy (N=71)
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 8 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 12 | 7
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 5 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 9 | 8
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3
Pain management (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphoma transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osmotic demyelination syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
8th nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breakthrough pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Creatinine renal clearance abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Tazemetostat 100 mg (N=6) | Phase 1: Tazemetostat 200 mg (N=3) | Phase 1: Tazemetostat 400 mg (N=3) | Phase 1: Tazemetostat 800 mg (N=14) | Phase 1: Tazemetostat 1600 mg (N=12) | Phase 1: Food Effect (All Patients) (N=13) | Phase 1: Tazemetostat 800 mg + Midazolam 2 mg (N=13) | Phase 2 Group 1: Tazemetostat in R/R FL With Mutant EZH2 (N=48) | Phase 2 Group 2: Tazemetostat in R/R FL With Wild-Type EZH2 (N=54) | Phase 2 Group 3: Tazemetostat in R/R DLBCL Monotherapy (N=163) | Phase 2 Group 4: Tazemetostat + Prednisolone in R/R DLBCL Combination Therapy (N=71)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 1 | 2 | 6 | 3 | 10 | 25 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 1 | 4 | 1 | 4 | 5 | 37 | 13
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 4 | 4 | 16 | 7
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 6 | 3 | 2 | 10 | 14 | 36 | 9
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 1 | 2 | 4 | 5 | 7 | 23 | 12
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2 | 3 | 3 | 5 | 3 | 14 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 2 | 0 | 1 | 11 | 10 | 28 | 11
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 8 | 5 | 12 | 12
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 8 | 2
Asthenia (General disorders) | 4 | 1 | 1 | 10 | 4 | 7 | 7 | 7 | 12 | 16 | 15
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 5 | 3 | 12 | 8
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 8 | 25 | 7
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 23 | 7
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 5 | 2 | 12 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 6 | 9 | 10 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 7 | 8 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 2 | 3 | 3 | 6 | 2 | 13 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 6 | 2 | 1 | 3 | 4 | 6 | 7 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 7 | 6 | 16 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 6 | 2 | 7 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 7 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 4 | 3 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2 | 2 | 2 | 3 | 6 | 7 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 7 | 11 | 32 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 7 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT01897571/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT01897571/SAP_001.pdf